CLINICAL TRIAL: NCT01239147
Title: Effect of Whole Grain Inclusion in the Diet on Abdominal Fat Regain After a Weight Loss Diet
Brief Title: Effects of Whole Grain on Weight Maintenance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cereal Partners Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2009.02.CPW / OP71709.UPC.CPW; NCT01848405 (obsolete NCT alias)
Record Dates: First submitted 2010-10-27; First posted 2010-11-11 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Abdominal Fat; Body Weight
Keywords: weight maintenance
MeSH Terms: conditions — Body Weight | interventions — Whole Grains

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole grain diet (Other)
  Interventions: Other: Diet rich in whole grain
- Refined grain diet (Other)
  Interventions: Other: Refined grain

INTERVENTIONS:
Other: Diet rich in whole grain — Ready-to-eat breakfast cereals and other cereal products, rich in whole grain
  Arms: Whole grain diet
Other: Refined grain — Ready-to-eat breakfast cereals and other cereal products, low in whole grain
  Arms: Refined grain diet

SUMMARY:
Epidemiological studies suggest that whole grain consumption affects measures of obesity including BMI, body fat tissue, and body weight. Most cross-sectional studies demonstrate rather consistently an inverse association between BMI and whole grain consumption. Furthermore, prospective cohort studies suggest that people with high whole grain consumption have less risk for body weight gain compared with low whole grain consumption.

The purpose of this study is to assess the effects of inclusion of whole grain in the diet on anthropometric measures, particularly abdominal fat regain after a weight loss diet.

It is anticipated that the short-term regain of abdominal fat after a weight loss diet is lower in volunteers consuming whole grain than in volunteers consuming refined grain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject, as determined by clinical examination, and medical history,
* Non-menopausal woman,
* BMI between 27 and 34 kg/m²
* Waist circumference > 80 cm.
* No diet within the last 3 months with weight loss or gain not more than 3kg.
* Non-smoking subject, or smoking less than 15 cigarettes/day since three months,
* Normal blood pressure (BP) and heart rate (HR) after 10 minutes in supine position. Individuals values out of the normal range can be accepted if judged clinically non relevant by the investigator.
* Laboratory parameters within the normal range of the laboratory (haematological, blood chemistry tests, urinalysis). Individual values out of the normal range can be accepted if judged clinically non relevant by the Investigator.
* Subject with a habitual low (< 16 g/day) intake of whole grain foods (from cereal food intake questionnaire),
* willing to eat breakfast cereals
* no intense physical activity,
* written consent to participate in the study,
* covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.
* registered in the national file of volunteers participating in biomedical research,
* Subject who has lost at least 6% initial body weight after the weight loss diet will be randomized to either the whole grain or the refined grain diet

Exclusion Criteria:

* Subject having a history of metabolic disease (i.e, diabetes),
* Subject suffering from chronic renal insufficiency
* Subject receiving a local or general treatment (i.e, prescription medications, over-the-counter medications, dietary supplements or herbal supplements) susceptible to interfere with the evaluation of the studied parameters and in particular weight (eg, appetite suppressants, slimming or treatment which could interfere with the metabolism and dietary behaviour),
* Subject with ongoing medication not stabilized since more than 3 months,
* Subject having had a general anaesthesia in the month preceding inclusion, or gastro-intestinal surgery at any time in his/her life, with the possible exception of appendectomy,
* Pregnant or breast-feeding subject (positive urinary pregnancy test),
* Subject in an exclusion period of a previous study or having participated in another clinical study in the last month,
* Use of laxatives, except in few occasions, if, in the opinion of the investigator, does not interfere with the optimal participation,
* Subject having received more than 4500 Euros in indemnity for participation in clinical studies in the last 12 months, including participation in the present study,
* Subject in a situation that, in the opinion of the investigator, could interfere with his optimal participation in the study or constitute a particular risk for the subject,
* Subject under any administrative or legal supervision.
* Subjects with known allergies to cereals

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 186 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Abdominal fat | 12 weeks
  Abdominal fat mass (DEXA)

SECONDARY OUTCOMES:
Body composition | 12 weeks
  Body composition (DEXA
body weight | 12 weeks
  body weight (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Yves DONAZZOLO, MD, MSc, Principal Investigator — Optimed Clinical Research
Locations (1):
- Optimed Clinical Research, Gières, France